CLINICAL TRIAL: NCT01057849
Title: Sequenced Atypical Antipsychotics Therapy With Intensive or Basic Psychosocial Intervention for First-episode Schizophrenia: An Effectiveness Study
Brief Title: Standard Comprehensive Intervention to Treat First-episode Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Xin Yu, Peking University Institute of Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007BAI17B04
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; first episode; atypical antipsychotics; psychosocial intervention; outcome; effectiveness
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Risperidone, Intensive (Experimental): risperidone and intensive psychosocial intervention
  Interventions: Drug: risperidone
- risperidone, basic (Active Comparator): risperidone and basic psychosocial support
  Interventions: Drug: risperidone
- olanzapine, intensive (Experimental): olanzapine and intensive psychosocial intervention
  Interventions: Drug: olanzapine
- olanzapine, basic (Active Comparator): olanzapine and basic psychosocial support
  Interventions: Drug: olanzapine
- aripiprazole, intensive (Experimental): aripiprazole and intensive psychosocial intervention
  Interventions: Drug: Aripiprazole
- aripiprazole, basiv (Active Comparator): aripiprazole and basic psychosocial support
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: risperidone — 3-6 mg per day
  Arms: Risperidone, Intensive; risperidone, basic
Drug: olanzapine — 5-20 mg per day
  Arms: olanzapine, basic; olanzapine, intensive
Drug: Aripiprazole — 10-30 mg per day
  Arms: aripiprazole, basiv; aripiprazole, intensive

SUMMARY:
Schizophrenia is not a curable but a treatable disease by antipsychotics. Kinds of atypical antipsychotics are widely used since 1990s' in China. Although their efficacy for acute phase are all better than typicals, individulized regimen of them for first-episode schizophrenia and their effectiveness in real naturalistic clinical settings still remain unclear. And those patients also need more comprehensive intervention such as psychosocial programs to improve their function. This protocol is to conduct a study in several sites of China to investigate the effectiveness of comprehensive intervention combining sequenced atypical antipsychotic therapy and intensive psychosocial intervention for first-episode schizophrenic patients. In addition, this protocol also aims at collecting such information as molecular genetics, neurochemical test, neucognitive performance and neuroimaging for outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenic patients diagnosed with DSM-IV criteria by SCID-I.
* age between 16-45 years old
* with disease course less than 3 years and during their first episode
* without receiving systematic antipsychotic treatment less than 1 month

Exclusion Criteria:

* organic disease or unstable physical diseases.
* brain trauma with loss of consciousness more than 1 hour
* current substance misuse (in 3 months) or any substance dependence.
* pregnant women.
* patients with severe suicidal imaginations or behavior.
* mental retardation
* contradict to the study drugs

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
the time the patients remain stable | 1 year

SECONDARY OUTCOMES:
Scoring of PANSS and PSP | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, M.D., Principal Investigator — Peking University Institute of Mental Health
Locations (6):
- China (6):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Institute of Mental Health, Haidian District, Beijing Municipality
  - Zhongnan University Xiangya Second Hospital, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Sichuan University Huaxi Hospital, Chengdu, Sichuan

REFERENCES:
- [Derived] Yin X, Zhou T, Huang B, Lu Z, Gao T, Guo X, Hu W, Ji Y, Wang X, Zheng Y, Yu X, Pu C. Trajectory analysis of BMI increase induced by second-generation antipsychotics in first-episode schizophrenia: a secondary analysis based on CNFEST***. Schizophrenia (Heidelb). 2025 Dec 4;12(1):7. doi: 10.1038/s41537-025-00710-1. PMID 41345405
- [Derived] Dai N, Huang B, Gao T, Zheng Y, Shi C, Pu C, Yu X. Initial attitudes toward a drug predict medication adherence in first-episode patients with schizophrenia: a 1-year prospective study in China. BMC Psychiatry. 2023 Dec 5;23(1):907. doi: 10.1186/s12888-023-05419-y. PMID 38053101
- [Derived] Cheng Z, Yuan Y, Han X, Yang L, Zeng X, Yang F, Lu Z, Wang C, Deng H, Zhao J, Yu X. Which Subgroup of First-Episode Schizophrenia Patients Can Remit During the First Year of Antipsychotic Treatment? Front Psychiatry. 2020 Jun 19;11:566. doi: 10.3389/fpsyt.2020.00566. eCollection 2020. PMID 32636771
- [Derived] Han X, Yuan YB, Yu X, Zhao JP, Wang CY, Lu Z, Yang FD, Dong H, Wu YF, Ungvari GS, Xiang YT, Chiu HF. The Chinese First-Episode Schizophrenia Trial: background and study design. East Asian Arch Psychiatry. 2014 Dec;24(4):169-73. PMID 25482837